CLINICAL TRIAL: NCT03264664
Title: An Open-Label, Multicenter, Phase 1 Study of E7386 in Subjects With Selected Advanced Neoplasms
Brief Title: Study of E7386 in Participants With Selected Advanced Neoplasms
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7386-G000-101; 2016-004881-25 (EudraCT Number)
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Advanced Neoplasms
Keywords: E7386; dose escalation; advanced or recurrent neoplasms; Hepatocellular carcinoma; HCC; CTNNB1 mutation
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular | interventions — E-7386

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E7386 BID (Experimental): E7386 will be administered as a single agent orally, initially twice daily (BID) continuously in 28 days treatment cycle. The dose will be escalated in cohorts of participants subject to safety data and the absence of DLTs. Based on the emerging data after completion of Dose Escalation Part, identifying MTD or RP2D, or after a decision is made to evaluate more than one potential RP2D level, a Dose Expansion Part will be initiated. Participants will continue to receive study treatment in extension phase until disease progression, development of unacceptable toxicity, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386

INTERVENTIONS:
Drug: E7386 — Oral immediate release tablets.

SUMMARY:
This study will be conducted to assess the safety/tolerability profile of E7386 as a single agent administered orally in participants with selected advanced or recurrent neoplasms and to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of E7386.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to (>=) 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy >=12 weeks
* Participant must have any of the following tumor types, confirmed by available histology or cytology records or current biopsy, that is advanced, nonresectable, recurrent since last antitumor therapy, in need of systemic treatment, and for which no alternative standard therapy exists:

  * Dose Escalation Part: Desmoid tumors, anaplastic thyroid cancer (ATC), endometrial cancer, melanoma, colorectal carcinoma (CRC), hepatocellular carcinoma (HCC), pancreatic cancer, prostate cancer, ovarian cancer, and head and neck cancer. Enrollment of additional tumor types will be discussed with the Sponsor and agreed on a case by case basis
  * Dose Expansion Part: HCC with CTNNB1 mutations as detected either in tumor tissue or circulating tumor DNA (ctDNA) by Sponsor-approved assay.

HCC participants must have:

i. Confirmed diagnosis of HCC ii. Barcelona Clinical Liver Cancer (BCLC) Stage C disease, or BCLC Stage B disease not amenable to local therapy.

* Participants must have accessible tumors to take biopsies from a pre-designated non target lesion for performance of correlative tissue studies. If the participant has only 1 measurable lesion and no other accessible lesion, the participant can be enrolled without a biopsy upon approval by the Sponsor
* Measurable disease meeting the following criteria:

  * At least 1 lesion of >=1.0 centimeter (cm) in the longest diameter for a non-lymph node or >=1.5 cm in the short-axis diameter for a lymph node that is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI)
  * Lesions that have had external beam radiotherapy (EBRT) or loco-regional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion
* Adequate renal function defined as serum creatinine less than or equal to (<=) 1.5*upper limit of normal (ULN), or for participants with serum creatinine greater than (>) 1.5*ULN, the calculated creatinine clearance >=30 milliliter per minute (mL/min) per the Cockcroft Gault formula (creatinine clearance >=40 mL/min for participants with HCC) is acceptable
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) >=1500/millimeters cubed (mm^3) (>=1.5*10^3/microliters [µl])
  * Platelets >=100,000/mm^3 (>=100*10^9/Liters [L]) (platelets >=75*10^9/L for participants with HCC)
  * Hemoglobin >=9.0 grams per deciliter (g/dL)
* Adequate liver function:

  * Total bilirubin <=1.5*ULN (<=2.0*ULN for participants with HCC)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=3*ULN (<=5*ULN if participant has liver metastases or participant with HCC)
* Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) <=1.5 (in the absence of therapeutic anticoagulation) (<=2.3 for participants with HCC)
* Normal serum calcium and potassium levels as per local laboratory reference ranges
* Serum magnesium greater than or equal to lower limit of normal as per local laboratory reference ranges
* Participants must agree to take vitamin D supplements continuously as per local institutional guidelines when 25-hydroxyvitamin D levels are less than 30 nanograms per milliliter (ng/mL)
* Willing and able to comply with all aspects of the protocol
* Provide written informed consent prior to any study-specific screening procedures
* Participants must have recovered from any previous anticancer therapy-related adverse events (AEs) to common terminology criteria for adverse events (CTCAE) v4.03 Grade equal to or less than (≤)1 (except for alopecia, ototoxicity, and Grade ≤2 peripheral neuropathy)

Exclusion Criteria:

* Other malignancy active within the previous 2 years except for basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast that has completed curative therapy
* Prior chemotherapy, immunotherapy (tumor vaccine, cytokine or growth factor given to control the cancer), or other anti-cancer therapy within less than 4 weeks before study drug administration; prior treatment with E7386
* Participants taking drugs, supplements, or foods that are known potent CYP3A4 inducers/inhibitors or sensitive substrates within less than 4 weeks before study drug administration
* Prior definitive radiation therapy within less than 4 weeks and prior palliative radiotherapy within less than 2 weeks before study drug administration. Radiopharmaceuticals (strontium, samarium) within less than 8 weeks before study drug administration
* Participants with brain or subdural metastases are not eligible, unless the metastases are asymptomatic and do not require treatment or have been adequately treated by local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks prior to study entry. Confirmation of radiographic stability must be done by comparing the brain scan (CT or MRI) performed during the Screening Period to a brain scan performed at least 4 weeks earlier (and following local therapy where applicable) using the same imaging modality as during the Screening Period. It is not the intention of this protocol to treat participants with active brain metastasis
* Known human immunodeficiency virus (HIV) infection
* (Dose escalation only) Active infection requiring therapy, including known positive tests for Hepatitis B surface antigen and hepatitis C virus (HCV) ribonucleic acid (RNA) (Dose expansion only) for participants with HCC: Has dual active HBV infection (HBV) and hepatitis C virus (HCV) infection at study entry.
* Major surgery within 4 weeks before the first dose of study drug or minor surgery within 1 week (participants must also have recovered from any surgery-related toxicities to CTCAE v4.03 Grade ≤1)
* Immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids (doses >10 milligrams [mg]/day prednisone or equivalent) within 2 weeks before study drug administration
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids except inhaled or intranasal corticosteroids (with minimal systemic absorption)
* Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (example, nausea, diarrhea, or vomiting) that might impair the bioavailability of E7386
* Prior receipt of bisphosphonate therapy for osteoporosis or symptomatic hypercalcemia or denosumab for osteoporosis
* Osteoporosis based on a T-score of <-2.5 at the left or right total hip, left or right femoral neck, or lumbar spine (L1-L4) as determined by dual energy x-ray absorptiometry (DXA) scan
* History of symptomatic vertebral fragility fracture or any fragility fracture of the hip, pelvis, wrist, or other location (defined as any fracture without a history of trauma or because of a fall from standing height or less)
* Moderate (25% or 40% decrease in the height of any vertebrae) or severe (>40% decrease in the height of any vertebra) morphometric vertebral fractures at baseline
* Bone metastases and one of the following:

  * Prior history of a recent (within 1 year prior to study entry) pathologic fracture
  * Lytic lesion requiring orthopedic intervention
  * Bone lesion requiring an impending orthopedic intervention
  * Lack of treatment with a bisphosphonate or denosumab (participants may be included if such treatment is started at least 14 days prior to Cycle 1 Day 1). Participants with previous solitary bone lesions controlled with radiotherapy are eligible
* Participants with known intolerance to study drug (or any of its excipients)
* Participants with a fasting serum β-C-terminal telopeptide (β-CTX) concentration of >1000 picograms (pg)/mL
* Participants with metabolic bone disease, such as hyperparathyroidism, Paget's disease, or osteomalacia
* Participants with a recent (within 6 months) history of or a newly diagnosed insufficiency fracture
* Use of other investigational drugs within 28 days or at least 5 half-lives (whichever is longer) before study drug administration.
* Use of any live vaccines (example, intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guérin (BCG), yellow fever, varicella, and TY21a typhoid vaccines) within 28 days prior to the first dose of study drug
* A prolonged QT/QT corrected (QTc) interval (QTc >450 milliseconds [ms]) as demonstrated by a repeated electrocardiogram (ECG). A history of risk factors for torsade de pointes (example, heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QT/QTc interval
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke, left ventricular ejection fraction (LVEF) <50% , cardiac arrhythmia requiring medical treatment (including oral anticoagulation) within 6 months prior to the first dose of study drug
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [β-hCG] test with a minimum sensitivity of 25 International Units per Liter [IU/L] or equivalent units of β-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
* Females of childbearing potential who:

  * Had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (example, true abstinence if it is their preferred and usual lifestyle [defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments], an intrauterine device, a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 4 weeks after study drug discontinuation
  * Are not currently abstinent, or do not agree to refrain from sexual activity during the study period and for 4 weeks after study drug discontinuation
  * Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study and for 4 weeks after study drug discontinuation (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [that is, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing])
* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (that is, not of childbearing potential or practicing highly effective contraception throughout the study period and for 4 weeks after study drug discontinuation). No sperm donation is allowed during the study period and for 4 weeks after study drug discontinuation
* Any other major illness, any history of a medical condition or a concomitant medical condition that, in the investigator's judgment, will substantially increase the risk associated with, or compromise the participant's participation in this study
* For participants with HCC, participants are excluded if:

  1. have a Child Pugh status of B and C.
  2. clear invasion to the bile duct or portal vein invasion of Vp4.
  3. symptomatic gastric or esophageal varices per Investigator's clinical judgement.
  4. history of hepatic encephalopathy within 6 months prior to starting study drug.
  5. (Dose Expansion only) cannot be evaluated by either triphasic liver CT or triphasic liver MRI because of allergy or other contraindication to both CT and MRI contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicities (DLTs) | Cycle 1 (28 days)
  DLTs are any of the pre-specified drug-related toxicities (any toxicities considered related to E7386) occurring during Cycle 1 as assessed by the investigator. DLTs will be assessed to determine the maximum tolerated dose.
Recommended Phase 2 Dose (RP2D) | Cycle 1 (28 days)
  RP2D will be selected based on an integrated evaluation of safety, tolerability, efficacy, pharmacokinetic (PK) data, and any available pharmacodynamic (PD) data for all dose levels or all available data according to pre-specified guidelines.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | From the date of first dose of study drug up to 28 days after administration of study drug (up to approximately 6 years and 10 months)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 6 years and 10 months
  ORR is defined as the proportion of participants achieving a best overall response of confirmed partial responses (PR) or complete response (CR), per Response Evaluation Criteria in Solid Tumors (RECIST 1.1). CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to less than (<) 10 millimeters (mm). PR is defined as at least a 30 percent (%) decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free Survival (PFS) | Up to approximately 6 years and 10 months
  PFS is defined as the time from the date of the first dose to the date of the first documentation of confirmed disease progression or death, whichever occurs first. Disease progression, per RECIST 1.1, is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Maximum Drug Concentration (Cmax) of E7386 | Cycle 1 Days 1 and 8: 0-12 hours postdose (Dose Escalation); Cycle 1-4 Day 1: 0-1 hours postdose (Dose Expansion) (each Cycle = 28 Days)
  Cmax is the maximum plasma concentration of a drug after administration.
Time to Reach the Maximum Concentration Following Drug Administration (tmax) of E7386 | Cycle 1 Days 1 and 8: 0-12 hours postdose (Dose Escalation); Cycle 1-4 Day 1: 0-1 hours postdose (Dose Expansion) (each Cycle = 28 Days)
  tmax is the time to reach maximum concentration following drug administration.
Area Under the Concentration Versus Time Curve (AUC) of E7386 | Cycle 1 Days 1 and 8: 0-12 hours postdose (Dose Escalation); Cycle 1-4 Day 1: 0-1 hours postdose (Dose Expansion) (each Cycle = 28 Days)
  AUC is a measure of actual body exposure to drug after administration of the drug.
Elimination Half-life (t1/2) of E7386 | Cycle 1 Days 1 and 8: 0-12 hours postdose (Dose Escalation); Cycle 1-4 Day 1: 0-1 hours postdose (Dose Expansion) (each Cycle = 28 Days)
  t1/2 is the time required for the concentration of the drug to reach half of its original value.
Apparent Total Body Clearance (CL/F) of E7386 | Cycle 1 Days 1 and 8: 0-12 hours postdose (Dose Escalation); Cycle 1-4 Day 1: 0-1 hours postdose (Dose Expansion) (each Cycle = 28 Days)
  CL/F is the volume of plasma cleared of drug per unit time.
Volume of Distribution (Vd) of E7386 | Cycle 1 Days 1 and 8: 0-12 hours postdose (Dose Escalation); Cycle 1-4 Day 1: 0-1 hours postdose (Dose Expansion) (each Cycle = 28 Days)
  Vd is the apparent volume in which a drug is distributed.
Renal Clearance (CLr) of E7386 | Cycle 1 Days 1 and 8: 0-24 hours postdose (Dose Escalation) (each Cycle = 28 Days)
Accumulation Ratio (R) of E7386 | Cycle 1 Days 1 and 8: 0-12 hours postdose (Dose Escalation); Cycle 1-4 Day 1: 0-1 hours postdose (Dose Expansion) (each Cycle = 28 Days)
  R indicates the extent to which drug accumulates.
Fraction Excreted (fe) of E7386 | Cycle 1 Days 1 and 8: 0-24 hours postdose (Dose Escalation) (each Cycle = 28 Days)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (5):
  - Mayo Clinic Comprehensive Caner, Phoenix, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Mayo Clinic Comprehensive Cancer, Jacksonville, Florida
  - Mayo Clinic Comprehensive Caner, Rochester, Minnesota
- United Kingdom (5):
  - The Beatson West of Scotland Cancer Centre, Glasgow, Lanarkshire
  - The Christie NHS Foundation Trust, Manchester, Lancashire
  - Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey
  - Royal Free London NHS Foundation Trust, Royal Free Hospital, London
  - Imperial College Healthcare NHS Trust, London